CLINICAL TRIAL: NCT00723177
Title: The Safety, Tolerability and Preliminary Efficacy of AV411, a Glial Activation Inhibitor, in Heroin Abusers Under Conditions of Morphine Maintenance and Withdrawal
Brief Title: Phase IIa Study of AV411, a Glial Activation Inhibitor, for Opioid Withdrawal
Acronym: AV411
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: #5725; P50DA009236 (NIH)
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Opioid-Related Disorders
Keywords: opioid withdrawal, analgesia
MeSH Terms: conditions — Opioid-Related Disorders; Agnosia | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): This group will receive placebo drug
  Interventions: Drug: Placebo (PCB)
- Low-dose AV411 (Experimental): This group will receive a low dose of AV411
  Interventions: Drug: AV411
- High-dose AV411 (Experimental): This group will receive a high dose of AV411
  Interventions: Drug: AV411

INTERVENTIONS:
Drug: AV411 — Low (20 mg), and high dose (40 mg) of AV411 will be administered orally twice a day (BID) for two consecutive weeks
  Other Names: ibudilast
  Arms: High-dose AV411; Low-dose AV411
Drug: Placebo (PCB) — Placebo drug will be administered orally twice a day (BID) for two consecutive weeks
  Other Names: PCB or 0 mg
  Arms: Placebo

SUMMARY:
Repeated use and/or abuse of opioid medications is generally associated with a characteristic withdrawal syndrome that develops after cessation of drug administration. The present study is designed to evaluate the effectiveness of AV411 to alter opioid-induced withdrawal symptoms.

DETAILED DESCRIPTION:
Opioid-induced cytokine release and glial activation has been proposed to directly contribute to the affective and physiological aspects of withdrawal. Furthermore, cytokine release following opioid administration has been hypothesized to be a limiting factor in both the duration and magnitude of opioid-induced analgesia. The two primary goals of our study are to assess AV411's ability to 1) reduce the opioid-withdrawal syndrome and 2) increase and prolong the analgesic effects of the mu-opioid agonist, oxycodone. To explore whether AV411 decreases opioid-induced glial cell activation, some participants assigned to the placebo and high dose AV411 groups (n = 6 for each dose condition) will be studied twice with [11C]PK11195, a positron emission tomography (PET) radiotracer used to measure the peripheral benzodiazepine receptor (PBR) in the human brain. The PBR is a receptor located on the mitochondria of the microglia and can be used to examine microglial activation in various brain regions.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 21 and 45
* Current dependence on heroin according to (Diagnostic and Statistical Manual) DSM-IV criteria
* Non-treatment seeking

Exclusion Criteria:

* Female participants who are currently pregnant or breastfeeding. Lack of effective birth control 10 days before Study Day 1 (15 days prior to the first PET scan)
* Self-reported use of methadone, buprenorphine, or levo-alpha-acetylmethadol (LAAM) in the past 14 days
* Participants who have a positive history of neurological illness (including epilepsy) or those who have received anti-convulsant therapy during the past 5 years
* Liver disease requiring medication or medical treatment, and/or aspartate or alanine aminotransferase levels greater than 3 times the upper limit of normal
* Gastrointestinal or renal disease that would significantly impair absorption, metabolism or excretion of study drug, or require medication or medical treatment
* Neurological or psychiatric disorders including psychosis, bipolar disorder, organic brain disease, any seizure history or other disorders that require treatment or that could make study compliance difficult
* Positive tuberculosis (PPD) TB skin test along with a clinical history and chest X-ray indicative of active tuberculosis. (Individuals who have a positive PPD test and have a negative chest X-ray, are not symptomatic for tuberculosis, and do not require anti-tuberculosis therapy will be eligible to participate. Participants will be asked if they ever tested positive for tuberculosis. If so, they will not be given a PPD and a chest X-ray and clinical history will be used for evaluation purposes).
* Presence or positive history of severe medical illness or any cardiovascular disease or heart abnormality, such as low hemoglobin (Hb < 13 g/dL in males, Hb < 11 g/dL in females), or BP > 150/90.
* Requirement for any of the following medications (current or within the past 4 weeks): psychotropics (including sedative/hypnotics, antidepressants, neuroleptics), anticonvulsants, antihypertensives, antiarrhythmics, or antiretroviral medications,. Participants on any current psychoactive prescription medications will be excluded.
* Current dependence (by DSM-IV criteria) on methadone, LAAM, or buprenorphine
* Participants for whom detoxification is not "clinically recommended" such as those with a significant history of overdose following detoxification
* Participation in an investigational drug study within the past 3 months
* Hypersensitivity to any of the medications used in this study
* Participants who are positive for HIV or chronic active hepatitis
* Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan, as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects" Shellock Frank G., Lippincott Williams & Wilkins Healthcare, Philadelphia, 2001.
* Lifetime exposure to radiation in the workplace, or participation in nuclear medicine procedures, including research protocols, in the past year
* Positive Allen Test indicating lack of collateral blood flow to hand
* History of Reynaud's syndrome

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, PhD, Principal Investigator — New York State Psychiatric Institute and Columbia University
Locations (1):
- New York State Psychiatric Institute/Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data have been published in a peer-reviewed journal.

REFERENCES:
- [Result] Cooper ZD, Johnson KW, Pavlicova M, Glass A, Vosburg SK, Sullivan MA, Manubay JM, Martinez DM, Jones JD, Saccone PA, Comer SD. The effects of ibudilast, a glial activation inhibitor, on opioid withdrawal symptoms in opioid-dependent volunteers. Addict Biol. 2016 Jul;21(4):895-903. doi: 10.1111/adb.12261. Epub 2015 May 14. PMID 25975386
- [Derived] Jacobsen JH, Watkins LR, Hutchinson MR. Discovery of a novel site of opioid action at the innate immune pattern-recognition receptor TLR4 and its role in addiction. Int Rev Neurobiol. 2014;118:129-63. doi: 10.1016/B978-0-12-801284-0.00006-3. PMID 25175864

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: This group received placebo AV411
  AV411: Placebo, low, and high dose of AV411 will be administered orally twice a day for two consecutive weeks
- Low-dose AV411: This group will receive a low dose of AV411
  AV411: Placebo, low, and high dose of AV411 will be administered orally twice a day for two consecutive weeks
- High-dose AV411: This group will receive a high dose of AV411
  AV411: Placebo, low, and high dose of AV411 will be administered orally twice a day for two consecutive weeks
Period: Overall Study
Arm/Group | Placebo | Low-dose AV411 | High-dose AV411
Started | 15 | 14 | 15
Completed | 10 | 10 | 10
Not Completed | 5 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: This group will receive placebo AV411
  AV411: Placebo, low, and high dose of AV411 will be administered orally BID for two consecutive weeks
- Low-dose AV411: This group will receive a low dose of AV411
  AV411: Placebo, low, and high dose of AV411 will be administered orally BID for two consecutive weeks
- High-dose AV411: This group will receive a high dose of AV411
  AV411: Placebo, low, and high dose of AV411 will be administered orally BID for two consecutive weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Low-dose AV411 | High-dose AV411 | Total
Number analyzed (Participants) | 15 | 14 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 15 | 44
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Year] | 39 (4.5) | 38 (5.3) | 38 (4.3) | 38 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 14 | 12 | 14 | 40
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Subjective Opioid Withdrawal Scale Score (SOWS)
Description: Measures severity of opioid withdrawal in opioid dependent populations (0-64). Larger values indicate more severe withdrawal.
Time Frame: Measured at the end of each two-week maintenance period (i.e., Placebo, Low AV411, High AV411).
Population: Only 30 of the total number of 44 enrolled completed the study .
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Low-dose AV411 | High-dose AV411
Number analyzed (Participants) | 10 | 10 | 10
units on a scale | 16 (4) | 4 (2) | 24 (10)

2. Secondary Outcome: The Effects of AV411 on the Analgesic Effects of Oxycodone.
Description: The McGill Pain Questionnaire (Melzack, 1987) was used to assess pain experience immediately following the immersion of the hand in 4 degree Celsius water. Scores were added across all 15 items to generate a sum score, which ranged between 15 and 60. Larger scores indicate greater pain levels.
Time Frame: Measured at the end of each AV411 of the three two-week maintenance periods
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low-dose AV411 | High-dose AV411
Number analyzed (Participants) | 10 | 10 | 10
units on a scale | 40 (5) | 42 (7) | 38 (5)

ADVERSE EVENTS:
Time Frame: We assessed for adverse events daily throughout the study and at 1 and 3 month follow-up time points. If a serious adverse events was experienced, it would have been reported to the appropriate oversight authorities within 24-48 hours.
Description: An adverse event (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. A serious adverse event is any AE that is: Fatal, Life-threatening, Requires or prolongs inpatient stay, Results in persistent or significant disability or incapacity.
Arm/Group | Placebo | Low-dose AV411 | High-dose AV411
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 2/14 | 5/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Low-dose AV411 (N=14) | High-dose AV411 (N=15)
GI upset and Constipation (Gastrointestinal disorders) | 3 (3) | 2 (4) | 2 (2)
Insomnia (Social circumstances) | 2 (3) | 2 (3) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No